CLINICAL TRIAL: NCT04983927
Title: An Open Label, Single-center, Retrospective, Pivotal Study to Evaluate the Efficacy of Clinical Decision Support System for Scoring of ASPECT Score Using Brain CT Images
Brief Title: Evaluation of Clinical Decision Support System for Scoring of ASPECT Score Using Brain CT Images
Status: Completed | Type: Observational
Sponsor: Heuron Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HR-cASP-01
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ischemic stroke positive: Patients diagnosed with acute ischemic stroke after a brain CT scan
  Interventions: Device: cASPECTS
- Ischemic stroke negative with other brain disease: Patients who has not been diagnosed with acute ischemic stroke after a brain CT scan, but has been diagnosed with other brain diseases.
  Interventions: Device: cASPECTS
- Ischemic stroke negative and no brain disease: Patients who has not been diagnosed with acute ischemic stroke after a brain CT scan and has not been diagnosed with other brain diseases.
  Interventions: Device: cASPECTS

INTERVENTIONS:
Device: cASPECTS — Clinical decision support system for scoring ASPECTS score

SUMMARY:
cASPECTS is a software that has been pre-learned based on ASPECTS Score of ischemic stroke patients using brain CT images, and clinical decision support system for scoring ASPECTS score by automatically analyzing brain CT images by assisting the medical team.

The specific aims of this study are to evaluate efficacy of cASPECTS for scoring ASPECTS Score compared to the sensitivity and specificity levels of human expert.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years old
* Brain CT acquired

Exclusion Criteria:

* Patients with ischemic stroke in posterior circulation
* Poor or incomplete brain CT image quality

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) Adults over 19 years old (2) Brain CT acquired are confirmed to be enrolled
Sampling Method: Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Differences between ASPECTS scores in golden standard and in cASPECTS | Within 4 weeks after collecting data
  Mean difference between ASPECTS scores calculated by human experts and ASPECTS scores calculated by cASPECTS

CONTACTS AND LOCATIONS:
Overall Officials: Daehan Choi, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, Namdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No